CLINICAL TRIAL: NCT01140204
Title: Restenosis Inhibition by Short-Term Exposure to Lipophilic Anti-proliferative Drugs Delivered by Angiographic Contrast Media
Brief Title: Short-Term Exposure to Lipophilic Anti-proliferative Drugs Delivered by Angiographic Contrast Media
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-325-02
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: stent; contrast media; paclitaxel; stent implantation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo control (Placebo Comparator): Contrast medium without Paclitaxel
  Interventions: Device: Implantation of a bare metal stent
- Iopromide Paclitaxel 0.85 mg (Active Comparator): Iopromide Paclitaxel 0.85 mg
  Interventions: Device: Implantation of a bare metal stent
- Iopromide Paclitaxel 4.27 mg (Active Comparator): Iopromide Paclitaxel 4.27 mg
  Interventions: Device: Implantation of a bare metal stent
- Iopromide Paclitaxel 8.54 mg (Active Comparator): Iopromide Paclitaxel 8.54 mg
  Interventions: Device: Implantation of a bare metal stent
- Iopromide Paclitaxel 17.08 mg (Active Comparator): Iopromide Paclitaxel 17.08 mg
  Interventions: Device: Implantation of a bare metal stent

INTERVENTIONS:
Device: Implantation of a bare metal stent — Bare Metal Stent

SUMMARY:
This was a randomized, placebo-controlled, multi-centre study, double-blind within each dose level, with four ascending dose levels to test the tolerability and safety of iopromide-paclitaxel in patients with de novo lesions in coronary arteries. Thirty-two patients were included into the trial, which were divided into four treatment groups. A total of four concentration levels of paclitaxel-iopromide concentrations were investigated. In each treatment group, six patients received iopromide-paclitaxel and two patients placebo (iopromide without paclitaxel). In each patient, the doses were adjusted individually as needed.

DETAILED DESCRIPTION:
Background: Non-stent-based immediate release formulations of paclitaxel have been shown to reduce in-stent restenosis in animal experiments and initial clinical trials. Paclitaxel dissolved in the angiographic contrast agent iopromide was well tolerated and inhibited neointimal proliferation in a dose-dependent manner after injection into porcine coronary arteries.

Methods: As a first step in entering clinical development, a phase I trial was performed using 4 ascending paclitaxel dose/concentration levels: samples of up to 100 ml of the contrast agent containing 10, 50, 100 or 200 μM paclitaxel were randomly administered to 6 adult patients each assigned to bare metal stent implantation for single de novo coronary artery lesions, while 8 patients treated with plain contrast medium served as controls. Safety variables and tolerability as well as angiographic parameters were assessed.

ELIGIBILITY:
Inclusion Criteria:

* male and postmenopausal female patients
* aged 18 years and older
* clinical evidence of stable or unstable angina, a positive functional test and a stentable de novo lesion in a native coronary artery
* diameter stenosis > 70% (visual estimate), lesion length < 25 mm, and a vessel diameter ≥ 2.5 mm.

Exclusion Criteria:

* acute myocardial infarction
* left ventricular ejection fraction of < 30%
* aorto-ostial lesion
* unprotected left main lesion or a bypass graft
* clear angiographic calcification in the target lesion
* visible thrombus proximal to the lesion
* chronic total occlusion
* platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* WBC <3,000 cells/mm3
* known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, abciximab, paclitaxel, stainless steel
* sensitivity to contrast media not amenable to adequate premedication
* medical illness (i.e. cancer, liver disease or congestive heart failure) associated with a life expectancy of less than two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-03; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Safety of intracoronary application | ca. 30 minutes (during intervention)
  * Continuous monitoring electrocardiogram (ECG)
  * Vital signs
  * Invasive measure of blood pressure
  * Lab variables: red blood count, white blood count, diff, creatinine kinase, creatinine kinase - muscle bound, creatinine
  * Cmax of paclitaxel in serum
  * 12-lead ECG
  * Adverse events

SECONDARY OUTCOMES:
Late lumen loss | 6 months
  Difference between angiographic in-stent minimum lumen diameter at 6 months follow-up and post-intervention
Restenosis rate | 6 months
  Defined as a diameter stenosis of ≥50% (assessed by quantitative coronary angiography) at any control angiography
Combined clinical endpoints (Major adverse cardiac events, MACE) | 6 months
  1. Abrupt and sub-abrupt closure
  2. Target lesion revascularization
  3. Myocardial infarction
  4. Death

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, MD, Principal Investigator — University Hospital, Saarland; Wolfgang Rutsch, MD, Principal Investigator — Charite Hospital, Berlin
Locations (2):
- Germany (2):
  - University Hospital of Saarland, Homburg/Saar, Saarland
  - Charite University Hospital, Berlin